CLINICAL TRIAL: NCT03126019
Title: A Phase 2, Multicenter, Open-Label Study of INCB050465, a PI3Kδ Inhibitor in Relapsed or Refractory Follicular Lymphoma (CITADEL-203)
Brief Title: A Study of INCB050465 in Relapsed or Refractory Follicular Lymphoma
Acronym: CITADEL-203
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCB 50465-203 (CITADEL-203); Parsaclisib (Other: Incyte Corporation); 2017-001624-22 (EudraCT Number)
Record Dates: First submitted 2017-04-20; First posted 2017-04-24 (Actual); Results first posted 2022-02-10 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Lymphoma
Keywords: Follicular lymphoma; non-Hodgkin lymphoma (NHL); phosphatidylinositol 3-kinase (PI3K) δ inhibitor
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Hereditary Sensory and Autonomic Neuropathies | interventions — parsaclisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A: Parsaclisib 20 mg QD for 8 Weeks Followed by 20 mg QW (Experimental): Participants received parsaclisib 20 mg once daily (QD) for 8 weeks followed by 20 mg once weekly (QW) for up to approximately 52 weeks.
  Interventions: Drug: Parsaclisib
- Treatment B: Parsaclisib 20 mg QD for 8 Weeks Followed by 2.5 mg QD (Experimental): Participants received parsaclisib 20 mg QD for 8 weeks followed by 2.5 mg QD for up to approximately 52 weeks.
  Interventions: Drug: Parsaclisib

INTERVENTIONS:
Drug: Parsaclisib — Parsaclisib tablets administered orally with water and without regard to food
  Other Names: INCB050465

SUMMARY:
The purpose of this study is to assess the objective response rate of parsaclisib treatment in participants with relapsed or refractory follicular lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* Histologically confirmed, relapsed or refractory, follicular B-cell non-Hodgkin lymphoma (NHL) (follicular lymphoma) Grade 1, 2, and 3a.
* Ineligible for hematopoietic stem cell transplant.
* Must have been treated with at least 2 prior systemic therapies.
* Radiographically measurable lymphadenopathy or extranodal lymphoid malignancy (defined as the presence of ≥ 1 lesion that measures > 1.5 cm in the longest dimension and ≥ 1.0 cm in the longest perpendicular dimension as assessed by computed tomography or magnetic resonance imaging.
* Must be willing to undergo an incisional, excisional, or core needle lymph node or tissue biopsy or provide a lymph node or tissue biopsy from the most recent available archival tissue.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.

Exclusion Criteria:

* Known histological transformation from indolent NHL to diffuse large B-cell lymphoma.
* History of central nervous system lymphoma (either primary or metastatic).
* Prior treatment with idelalisib, other selective phosphatidylinositol 3-kinase delta (PI3Kδ) inhibitors, or a pan-PI3K inhibitor.
* Prior treatment with a Bruton's tyrosine kinase inhibitor (eg, ibrutinib).
* Allogeneic stem cell transplant within the last 6 months, or autologous stem cell transplant within the last 3 months before the date of study treatment administration.
* Active graft-versus-host disease.
* Participants positive for hepatitis B surface antigen or hepatitis B core antibody will be eligible if they are negative for hepatitis B virus-deoxyribonucleic acid (HBV-DNA). Participants positive for anti-hepatitis C virus (HCV) antibody will be eligible if they are negative for HCV-ribonucleic acid (RNA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2024-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Zheng, MD, PhD, Study Director — Incyte Corporation
Locations (83):
- United States (22):
  - Arizona Oncology Associates - Biltmore Cancer Center, Phoenix, Arizona
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Synergy Hematology and Oncology Medical Associates, Los Angeles, California
  - St. Joseph Heritage Healthcare, Santa Rosa, California
  - American Institute of Research Corporate Office, Whittier, California
  - Cancer Center of Central Connecticut, Southington, Connecticut
  - Florida Cancer Specialists & Research Institute, Fort Myers, Florida
  - Asclepes Research Centers, Spring Hill, Florida
  - Clinical Trials of Swla Llc, Lake Charles, Louisiana
  - Saint Agnes Hospital, Baltimore, Maryland
  - Barbara Ann Karmanos Cancer Hospital, Detroit, Michigan
  - Hattiesburg Clinic Hematology, Hattiesburg, Mississippi
  - Saint Luke'S Hospital, Kansas City, Missouri
  - Sarah Cannon Research Institute, Kansas City, Missouri
  - Clinical Research Alliance, Inc., New Hyde Park, New York
  - Duke University Medical Center, Durham, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Charleston Hematology Oncology Associates Pa, Charleston, South Carolina
  - Tennessee Oncology, Nashville, Tennessee
  - Renovatio Clinical Consultants Llc, Spring, Texas
  - University of Washington, Seattle, Washington
- Australia (3):
  - Western Health, St Albans, Victoria
  - Border Medical Oncology, Wodonga, Victoria
  - St Vincent'S Hospital Sydney, Darlinghurst
- Canada (3):
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - Santa Cabrini Hospital, Montreal, Quebec
- Czechia (5):
  - University Hospital Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Ostrava, Ostrava
  - University Hospital Kralovkse Vinohrady, Prague
  - Univerzita Karlova V Praze 1. Lekarska Fakulta, Prague
  - Fakultni Nemocnice V Motole, Prague
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Odense Universitetshospital (Ouh) (Odense University Hospital), Odense C
- Germany (4):
  - Bag Arnoldstr. Dresden, Dresden
  - University Medical Center Freiburg, Freiburg im Breisgau
  - Universitatsmedizin Der Johannes Gutenberg-Universitat Mainz Iii, Mainz
  - University Hospital Mannheim, Mannheim
- Hungary (4):
  - Semmelweis Egyetem, Budapest
  - National Institute of Oncology, Budapest
  - University of Debrecen, Debrecen
  - Somogy Medyei Kaposi Mor Oktato Korhaz, Kaposvár
- Israel (5):
  - Hillel Yafe Medical Center (Hymc), Hadera
  - Rambam Medical Center, Haifa
  - Laniado Hospital Hematology, Netanya
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (14):
  - Irccs Centro Di Riferimento Oncologico, Aviano
  - Istituto Tumori Giovanni Paolo Ii Irccs Ospedale Oncologico Bari, Bari
  - University of Bologna, Bologna
  - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori, Meldola
  - Ospedale San Raffaele, Milan
  - Fondazione Irccs Istituto Nazionale Dei Tumori, Milan
  - A.O.U. Di Modena - Policlinico, Modena
  - A.O.U. Federico Ii, Napoli
  - Aou Maggiore Della Carita, Novara
  - Ospedali Riuniti Villa Sofia Cervello, Palermo
  - Sapienza University, Rome
  - I.R.C.C.S. Casa Sollievo Della Sofferenza, San Giovanni Rotondo
  - Aou Citta Della Salute E Della Scienza Di Torino, Torino
  - San Bartolo Hospital, Vicenza
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Pratia McM Krakow, Krakow
  - State Hospital Opole, Opole
  - Institute of Hematology and Transfusion Medicine, Warsaw
  - Centrum Onkologii-Instytut Im. Marii Sklodowskiej-Curie, Warsaw
- Spain (11):
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital General Universitari Vall D Hebron, Barcelona
  - Hgu Gregorio Maranon, Madrid
  - Md Anderson Cancer Centre Madrid, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario de La Paz, Madrid
  - Hospital Universitario Hm Sanchinarro, Madrid
  - Hospital Universitario Quironsalud Madrid, Madrid
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen Del Rocio, Seville
- Karolinska University Hospital, Huddinge, Stockholm, Sweden
- United Kingdom (4):
  - Birmingham Heartlands Hospital, Birmingham
  - Northwick Park Hospital, London
  - Royal Hallamshire Hospital, Sheffield
  - The Royal Marsden Nhs Foundation Trust - Chelsea, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 44 investigative sites in the United States, Italy, Spain, Great Britain, Czech Republic, Hungary, Canada, Denmark, Germany, Israel, Poland, and Sweden
Pre-assignment Details: A total of 126 participants with relapsed or refractory follicular lymphoma were enrolled in the study and assigned to one of two treatment groups: Treatment A or Treatment B to receive parsaclisib.
Groups:
- Treatment A: Parsaclisib 20 mg QD for 8 Weeks Followed by 20 mg QW: Participants received parsaclisib 20 milligrams (mg) once daily (QD) for 8 weeks followed by 20 mg once weekly (QW) for up to approximately 52 weeks.
Period: Overall Study
Arm/Group | Treatment A: Parsaclisib 20 mg QD for 8 Weeks Followed by 20 mg QW | Treatment B: Parsaclisib 20 mg QD for 8 Weeks Followed by 2.5 mg QD
Started | 23 | 103
Completed | 14 | 50
Not Completed | 9 | 53
Not completed — Death | 5 | 27
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 1 | 9
Not completed — Physician Decision | 1 | 0
Not completed — Transitioned to Rollover Study | 0 | 11
Not completed — Did Not Return to Site for Care | 0 | 1
Not completed — Site Closed | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all participants enrolled in the study who received at least 1 dose of parsaclisib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A: Parsaclisib 20 mg QD for 8 Weeks Followed by 20 mg QW | Treatment B: Parsaclisib 20 mg QD for 8 Weeks Followed by 2.5 mg QD | Total
Number analyzed (Participants) | 23 | 103 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (11.56) | 67.0 (10.68) | 66.5 (10.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 45 | 56
  Male | 12 | 58 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 6 | 7
  Not Hispanic or Latino | 19 | 90 | 109
  Unknown or Not Reported | 3 | 7 | 10
Race Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  Black/ African- American | 1 | 6 | 7
  White/ Caucasian | 21 | 92 | 113
  Unavailable or Unknown | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate With Parsaclisib Based on Lugano Classification Response Criteria
Description: ORR=percentage of participants with complete response(CR) or partial response(PR) per revised response criteria for lymphomas,determined by independent review committee(IRC).Criteria for CR:1.Target nodes/nodal masses of lymph nodes,extralymphatic sites regressed to≤1.5cm in longest dimension transverse diameter of lesion(LDi);2.Absence of non-measured lesion;3.Organ enlargement regressed to normal;4.No new lesions;5.Normal bone marrow morphology;if indeterminate,immunohistochemistry negative.Criteria for PR:1.Lymph nodes,extralymphatic sites- ≥50%decrease in sum of product of perpendicular diameters for multiple lesions(SPD)of up to 6 target measurable nodes,extranodal sites;if lesion is too small to measure on computed tomography(CT),assign5mm×5mm as default;if no longer visible,0×0mm.Node>5mm×5mm but smaller than normal,use actual measurement.2.Absent/regressed non-measured lesions,no increase.3.Organ enlargement-Spleen regressed by>50%in length beyond normal.4.No new lesions.
Time Frame: Up to approximately 148 weeks
Population: Full Analysis Set: all participants enrolled in the study who received at least 1 dose of parsaclisib
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment A: Parsaclisib 20 mg QD for 8 Weeks Followed by 20 mg QW | Treatment B: Parsaclisib 20 mg QD for 8 Weeks Followed by 2.5 mg QD
Number analyzed (Participants) | 23 | 103
percentage of participants | 65.2 [42.7 to 83.6] | 77.7 [68.4 to 85.3]

2. Secondary Outcome: Complete Response Rate With Parsaclisib Based on Lugano Classification Response Criteria
Description: CRR was defined as the percentage of participants with a CR as defined by revised response criteria for lymphomas as determined by an IRC. The criteria for CR included: 1. Target nodes/nodal masses of lymph nodes and extralymphatic sites must regress to ≤ 1.5 cm in LDi; 2. Absence of non-measured lesion; 3. Organ enlargement regressed to normal; 4. No new lesions; 5. Bone marrow must be normal by morphology; if indeterminate, immunohistochemistry negative.
Time Frame: Up to 1193 days
Population: Full Analysis Set: all participants enrolled in the study who received at least 1 dose of parsaclisib
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment A: Parsaclisib 20 mg QD for 8 Weeks Followed by 20 mg QW | Treatment B: Parsaclisib 20 mg QD for 8 Weeks Followed by 2.5 mg QD
Number analyzed (Participants) | 23 | 103
percentage of participants | 17.4 [5.0 to 38.8] | 22.3 [14.7 to 31.6]

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR=time from first documented evidence of CR or PR until disease progression or death from any cause among participants who achieve an objective response as determined by IRC. Criteria for CR: 1.Target nodes/nodal masses of lymph nodes and extralymphatic sites must regress to ≤ 1.5 cm in LDi; 2. Absence of non-measured lesion; 3.Organ enlargement regressed to normal; 4.No new lesions; 5.Bone marrow must be normal by morphology; if indeterminate, immunohistochemistry negative. The criteria for PR included: 1.Lymph nodes and extralymphatic sites- a. ≥50% decrease in SPD of up to 6 target measurable nodes and extranodal sites; b. when a lesion is too small to measure on CT, assign 5 mm×5 mm as the default; c.when no longer visible, 0×0 mm. For a node >5 mm×5 mm but smaller than normal, use actual measurement. 2.Non-measured lesions- Absent/regressed, but no increase. 3. Organ enlargement-Spleen must have regressed by >50% in length beyond normal. 4.No new lesions.
Time Frame: Up to 1193 days
Population: Full Analysis Set: all participants enrolled in the study who received at least 1 dose of parsaclisib. Only participants with objective response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment A: Parsaclisib 20 mg QD for 8 Weeks Followed by 20 mg QW | Treatment B: Parsaclisib 20 mg QD for 8 Weeks Followed by 2.5 mg QD
Number analyzed (Participants) | 15 | 81
months | 14.06 [3.19 to NA] — The upper limit of the 95% confidence interval (CI) was not estimable due to the low number of participants with events of response. | 14.72 [11.76 to 25.72]

4. Secondary Outcome: Progression-free Survival (PFS) With Parsaclisib
Description: PFS was defined as the time from the date of the first dose of study treatment until the earliest date of disease progression, as determined by radiographic disease assessment provided by an IRC, or death from any cause.
Time Frame: Up to 1193 days
Population: Full Analysis Set: all participants enrolled in the study who received at least 1 dose of parsaclisib
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment A: Parsaclisib 20 mg QD for 8 Weeks Followed by 20 mg QW | Treatment B: Parsaclisib 20 mg QD for 8 Weeks Followed by 2.5 mg QD
Number analyzed (Participants) | 23 | 103
months | 19.32 [8.31 to 33.15] | 14.03 [11.07 to 20.07]

5. Secondary Outcome: Overall Survival (OS) With Parsaclisib
Description: OS was defined as the time from the date of the first dose of study treatment until death from any cause.
Time Frame: Up to 1193 days
Population: Full Analysis Set: all participants enrolled in the study who received at least 1 dose of parsaclisib
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment A: Parsaclisib 20 mg QD for 8 Weeks Followed by 20 mg QW | Treatment B: Parsaclisib 20 mg QD for 8 Weeks Followed by 2.5 mg QD
Number analyzed (Participants) | 23 | 103
months | NA [35.48 to NA] — The median and the upper limit of the 95% CI were not estimable due to the low number of participants with events. | NA [NA to NA] — The median and the lower and upper limits of the 95% CI were not estimable due to the low number of participants with events.

6. Secondary Outcome: Best Percent Change From Baseline in Target Lesion Size
Description: Target lesion size is measured by the sum of the product of diameters of all target lesion sizes and is determined by the IRC. The best percent change from Baseline is defined as the largest decrease, or smallest increase (if no decrease available), from Baseline in target lesion sizes on/before new (next-line) anti-lymphoma therapy during the study. Baseline is the last non-missing measurement obtained before the first administration of study drug. A negative percent change from Baseline indicates improvement.
Time Frame: Up to 1193 days
Population: Full Analysis Set: all participants enrolled in the study who received at least 1 dose of parsaclisib. The overall number of participants analyzed is the number of participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: percent change in lesion size
Arm/Group | Treatment A: Parsaclisib 20 mg QD for 8 Weeks Followed by 20 mg QW | Treatment B: Parsaclisib 20 mg QD for 8 Weeks Followed by 2.5 mg QD
Number analyzed (Participants) | 20 | 98
percent change in lesion size | -72.90 (21.782) | -72.77 (31.972)

7. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence associated with use of a drug in humans, whether or not considered drug related, that occurs after a participant provides informed consent. TEAE is any AE either reported for first time or worsening of a pre-existing event after first dose of study drug and within 30 days of last administration of study drug regardless of starting new anti-lymphoma therapy. SAE is any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, leads to a congenital anomaly/birth defect or is considered to be an important medical event that may not result in death, be immediately life-threatening, or require hospitalization but may be considered serious when, based on appropriate medical judgment, the event may jeopardize the participant or may require medical or surgical intervention.
Time Frame: up to approximately 1992 days
Population: Safety Population: all participants enrolled in the study who received at least 1 dose of parsaclisib
Measure: Number; unit: percentage of participants
Arm/Group | Treatment A: Parsaclisib 20 mg QD for 8 Weeks Followed by 20 mg QW | Treatment B: Parsaclisib 20 mg QD for 8 Weeks Followed by 2.5 mg QD
Number analyzed (Participants) | 23 | 103
percentage of participants
  TEAEs | 100.0 | 99.0
  SAEs | 52.2 | 53.4

ADVERSE EVENTS:
Time Frame: up to approximately 1992 days
Description: Adverse events have been reported for members of the Safety Population, comprised of all participants enrolled in the study who received at least 1 dose of parsaclisib.
Arm/Group | Treatment A: Parsaclisib 20 mg QD for 8 Weeks Followed by 20 mg QW | Treatment B: Parsaclisib 20 mg QD for 8 Weeks Followed by 2.5 mg QD
All-Cause Mortality (participants affected / at risk) | 5/23 | 27/103
Serious Adverse Events (participants affected / at risk) | 12/23 | 55/103
Other Adverse Events (participants affected / at risk) | 22/23 | 94/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A: Parsaclisib 20 mg QD for 8 Weeks Followed by 20 mg QW (N=23) | Treatment B: Parsaclisib 20 mg QD for 8 Weeks Followed by 2.5 mg QD (N=103)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Autoimmune arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 1 (1)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Campylobacter colitis (Infections and infestations) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 8 (8)
Colitis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus colitis (Infections and infestations) | 1 (1) | 1 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Desmoplastic mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 10 (11)
Disease progression (General disorders) | 0 (0) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Parotid gland enlargement (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (6)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 3 (4)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Stomal hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A: Parsaclisib 20 mg QD for 8 Weeks Followed by 20 mg QW (N=23) | Treatment B: Parsaclisib 20 mg QD for 8 Weeks Followed by 2.5 mg QD (N=103)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 9 (12)
Alanine aminotransferase increased (Investigations) | 1 (1) | 7 (11)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 16 (17)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 8 (9)
Asthenia (General disorders) | 2 (2) | 14 (17)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 9 (9)
C-reactive protein increased (Investigations) | 2 (2) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1) | 10 (12)
Constipation (Gastrointestinal disorders) | 1 (1) | 11 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 28 (30)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 12 (13)
Diarrhoea (Gastrointestinal disorders) | 3 (5) | 45 (75)
Dizziness (Nervous system disorders) | 1 (1) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 8 (10)
Extrasystoles (Cardiac disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 3 (3) | 21 (23)
Headache (Nervous system disorders) | 1 (1) | 14 (14)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3) | 7 (8)
Hypertension (Vascular disorders) | 0 (0) | 12 (13)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 13 (16)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 10 (12)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Nausea (Gastrointestinal disorders) | 8 (8) | 28 (34)
Neutropenia (Blood and lymphatic system disorders) | 2 (4) | 16 (21)
Oedema peripheral (General disorders) | 1 (1) | 10 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 8 (8)
Peripheral swelling (General disorders) | 2 (2) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (6) | 3 (5)
Pyrexia (General disorders) | 2 (2) | 20 (26)
Rash (Skin and subcutaneous tissue disorders) | 6 (8) | 15 (18)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 7 (8)
Urinary tract infection (Infections and infestations) | 3 (3) | 6 (6)
Vomiting (Gastrointestinal disorders) | 3 (4) | 9 (10)
Weight decreased (Investigations) | 0 (0) | 6 (6)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2019-12-23): https://cdn.clinicaltrials.gov/large-docs/19/NCT03126019/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/19/NCT03126019/SAP_001.pdf